CLINICAL TRIAL: NCT05379842
Title: Educational Strategy on a Vulnerable Population to Improve Cardiovascular Health and Mitigate Food Insecurity Through a Sustainable Health Literacy Program
Brief Title: Educational Strategy on a Vulnerable Population to Improve Cardiovascular Health and Food Insecurity
Acronym: E-DUCASS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI20/01413
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Health; Food Insecurity; Healthy Lifestyle; Vulnerable Population
Keywords: Food insecurity; Educational program; Health Literacy; Cardiovascular Health; E-learning; Healthy Planetary Food
MeSH Terms: interventions — Health Literacy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1- Non-intervention (No Intervention): Non-posterior intervention after randomization
- 2- Traditional advanced intervention model (Active Comparator): Motivational workshops, every 3 months and with limited cost
  Interventions: Other: Education on a healthy lifestyle and health literacy
- 3- E-learning advanced intervention model (Active Comparator): Educational workshops, every 15 days, with videos -YouTube channel or WhatsApp/text message
  Interventions: Other: Education on a healthy lifestyle and health literacy

INTERVENTIONS:
Other: Education on a healthy lifestyle and health literacy — Traditional motivational face-to-face workshops with lifestyle (nutritional, physical activity, sleep) advice every 3 months
  Arms: 2- Traditional advanced intervention model
Other: Education on a healthy lifestyle and health literacy — E-learning and digital (with videos -YouTube channel or WhatsApp/text message) educational workshops with lifestyle (nutritional, physical activity, sleep) advice every 15 days
  Arms: 3- E-learning advanced intervention model

SUMMARY:
The purpose of this study is to demonstrate that an educational program on a healthy lifestyle which increases health literacy could improve long-term health and mitigate food insecurity.

DETAILED DESCRIPTION:
A 24-month randomized clinical trial involving vulnerable families (460 participants) at risk of food insecurity to improve cardiovascular health, with an initial basic training workshop followed by randomization into three groups: 1. No further intervention; 2. A traditional advanced intervention model every three months; and 3. E-learning advanced intervention model every 15 days with YouTube videos and WhatsApp messages.

Primary objective:

- Improve cardiovascular health measured by Life's Simple 7, American Heart Association

Secondary objective

* Demonstrate whether the intervention improves the food safety score measured according to FAO
* Study which of the two models of advanced intervention, face-to-face or virtual, improves cardiovascular and food health literacy in the study population.

This project aims to transfer and offer to society this virtual educational strategy as a tool to improve cardiovascular health in other vulnerable populations, in a scientific, efficient, safe, and sustainable way.

ELIGIBILITY:
Inclusion Criteria:

* Participants from the general population without disabling diseases or whose severity implies a life expectancy of less than five years
* Informed Consent

Exclusion Criteria:

* Age less than 12 years or equal to or greater than 80 years, with a life expectancy, not less than 5 years.
* Patients with established cardiovascular disease
* Patients with limitations to follow the protocol
* Serious or difficult-to-control risk factors: Patients with hypertension and diabetes with organic involvement that limits their survival and disabling clinical manifestations of cerebral arteriosclerosis will be excluded.
* Chronic diseases not related to coronary risk: severe psychiatric diseases, chronic processes requiring treatment such as chronic renal failure, chronic liver disease, neoplasms undergoing treatment, severe and very severe chronic obstructive pulmonary disease, endocrinopathies susceptible to decompensation, and digestive tract diseases.
* Participants in other clinical trials at screening or within 30 days prior to start.
* Excessive alcohol and drug abuse
* Pregnant or lactating women.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Health | 24 months
  Improve cardiovascular health measured by Life's Simple 7 (LS7) score. LS7 score is composed of seven domains (diet, physical activity, body mass index, smoking, blood pressure, total cholesterol and fasting blood glucose). Each of seven domains were ranged from 0 poor to 2 ideal. The total score of LS7 ranged from 0-14 with higher scores indicating better cardiovascular health.
Food insecurity | 24 months
  Improve food insecurity measured by The Food Insecurity Experience Scale Survey Module (FIES-SM) from Food and Agriculture Organization of the United Nations. FIES-SM is composed of eight questions with dichotomous no (0 points)/ yes (1 point) responses. The final score ranged from 0 (no insecurity food) to 8 (worst insecurity food).

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Pérez Martínez, PhD MD, Principal Investigator — Maimonides Institute for Biomedical Research in Cordoba (IMIBIC), Reina Sofia University Hospital
Locations (1):
- Reina Sofia University Hospital, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romero-Cabrera, Juan L.; de-Castro-Burón, Isabel; Yubero-Serrano, Elena; Díaz-Cáceres, Alberto; Serrán-Jiménez, Alejandro; Arenas-Montes, Javier; Alcalá-Díaz, Juan F.; Ortiz-Morales, Ana; Pérez-Martínez, Pablo. (2022). Educational strategy to improve cardiovascular health and mitigate food insecurity: Rationale for the E-DUCASS program. Spanish Journal of Medicine. 2. 10.24875/SJMED.21000025.
- [Derived] Porras-Perez E, Romero-Cabrera JL, Diaz-Caceres A, Serran-Jimenez A, Arenas-Montes J, Pena-Orihuela PJ, De-Castro-Buron I, Garcia-Rios A, Torres-Pena JD, Malagon MM, Delgado-Lista J, Ordovas JM, Yubero-Serrano EM, Perez-Martinez P. Food Insecurity and Its Cardiovascular Implications in Underresourced Communities. J Am Heart Assoc. 2025 Mar 18;14(6):e037457. doi: 10.1161/JAHA.124.037457. Epub 2025 Mar 13. PMID 40082777